CLINICAL TRIAL: NCT02110472
Title: Prospective, Non-randomized, Unmasked, Multicenter Clinical Investigation of the Presbia Flexivue Microlens™ for the Improvement of Near Vision in Emmetropic Presbyopes
Brief Title: Investigation of the Presbia Flexivue Microlens™
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PresbiBio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CLP-12-001
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Presbyopia
Keywords: Emmetropic presbyopes; Presbyopic
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Presbia Flexivue Microlens Corneal Inlay (Other): Presbia Flexivue Microlens implanted in corneal pocket in nondominant eye
  Interventions: Device: Corneal inlay

INTERVENTIONS:
Device: Corneal inlay — Presbia Flexivue Microlens implantation in corneal pocket created in nondominant eyes of emmetropic presbyopes.
  Other Names: Presbia Flexivue Microlens; Presbia Microlens

SUMMARY:
The Presbia Flexivue Microlens is a corneal inlay.

DETAILED DESCRIPTION:
Presbyopia is a multifactorial physiological aging mechanism that leads to a progressive functional loss of near vision. In addition to the use of reading glasses for presbyopia, a wide variety of procedures have been investigated by ophthalmologists to correct this refractive error. Cornea laser surgery with multifocal patterns or monovision approaches were developed including LASIK, PresbyLASIK, photorefractive keratectomy (PRK), laser epithelial keratomileusis (LASEK), thin-flap femto-LASIK or sub-Bowman's keratomileusis (SBK). Conductive keratoplasty (CK), clear lens extraction or cataract surgery using multifocal, pseudo-accommodative intraocular lenses (IOLs) or monovision monofocal IOLs are also some of the techniques that have been used for the treatment of presbyopia.

Corneal laser surgery and CK are minimally invasive methods, but they provoke irreversible changes of the corneal anatomy, whereas scleral surgery and clear lens extraction are more invasive techniques. The necessity to develop a minimally invasive, reversible, and safe surgical technique with an easy learning curve for patients between 45 and 60 years, led to the development of refractive intracorneal lenses (inlays) (such as the AcuFocus, Inc. KAMRA™, ReVision Optics® PresbyLens®, and the Presbia Flexivue Microlens™) placed inside the corneal stroma. These inlays are refractive lenses that have a central zone free of refractive power and a peripheral zone with a standard positive refractive power. These inlays are inserted inside the corneal stroma of the non-dominant eye, generally offering two different focal points, one for the far vision and a different for the near vision respectively. The pocket of the cornea is created using a laser (details to be provided later in this protocol).

The Presbia Flexivue Microlens is intended to improve near vision and decrease dependence on reading glasses in presbyopic adults who are tolerant of monovision (as evaluated by participation in a monovision tolerance trial (5 to 7 days minimum)), who require a reading add of +1.50 D to +3.50 D, who have MRSE between +1.00 D and 0.75 D with no more than 0.75 D of refractive cylinder, and who have stable MRSE within 0.50 D over the past 12 months.

Objective: The primary objective of this study is to evaluate the safety and effectiveness of the Presbia Flexivue Microlens™ (hereinafter referred to as the "Microlens") implanted in presbyopes for improvement of near vision.

Investigational Plan: This is a prospective, non-randomized, unmasked, multicenter clinical investigation. A total of 412 subjects at up to 11 investigational sites in the United States will undergo insertion of the Microlens in non-dominant eyes, and will be followed through 36 months postoperative (assuming an estimated 10% per year lost to follow-up). Each site will contribute a targeted minimum of 20 treated subjects, but no more than 25% of the total subjects treated in the study. Data on a minimum of 300 subjects with 24 month data will be submitted as part of the Premarket Approval; all subjects will be followed through 36 months postoperative. Subjects from outside the United States will not be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be emmetropes with presbyopia, between ≥ 45 years and ≤ 60 years of age at time of eligibility visit.
* Subjects must need a reading add of +1.50 D to +3.50 D.
* Subjects must have uncorrected near visual acuity of 20/50 or worse.
* Subjects must have near visual acuity correctable to 20/20 or better in each eye.
* Subjects must have distance visual acuity correctable to 20/25 or better in each eye.
* Subjects must have a preoperative spherical equivalent of +1.00 D to -0.75 D with no more than 0.75 D of refractive cylinder as determined by cycloplegic refraction in each eye.
* Subjects must have a photopic pupil size of > 1.6 mm in the eye to be implanted.

Exclusion Criteria:

* Subjects in whom the non-dominant eye cannot be determined using one of the methods identified in the test of ocular dominance.
* Subjects who do not complete the monovision tolerance trial (minimum of 5 to 7 days).
* Subjects who report that they were not completely satisfied with their vision during the monovision tolerance trial.
* Subjects who report that they experienced debilitating or significant visual symptoms such as halos, glare, double vision, etc. during the monovision tolerance trial.
* Subjects with a difference of ≥ 1.00 D between the spherical equivalent manifest refraction and the spherical equivalent cycloplegic refraction.
* Subject with a preferred near working distance of < 35 cm or > 45 cm.
* Subjects with corneal thickness < 500 microns in the eye to be implanted.
* Subjects with clinically significant anterior segment pathology, including cataracts, in either eye.
* Subjects with residual, recurrent, active ocular or uncontrolled eyelid disease or any progressive corneal abnormalities (including endothelial dystrophy, guttata in the central cornea, etc.) in the eye to be treated.
* Subjects with keratoconus (or keratoconus suspect), amblyopia, recurrent erosion syndrome or corneal dystrophy in the eye to be treated.
* Subjects with a history of chronic dry eye not controlled on therapy or with superficial punctuate keratitis (SPK) grade > II (i.e., greater than mild) based on Oxford Grading Scale in the eye to be treated.
* Subjects with abnormal corneal mires on topography maps of the eye to be treated.
* Subjects who require canthotomy to generate a corneal tunnel in the eye to be treated.
* Subjects with progressive retinal pathology with a reasonable chance of causing a reduction in BCVA from preoperative in the eye to be treated.
* Subjects who have undergone previous intraocular or corneal surgery including cataract and refractive surgery (e.g., LASIK surgery) in either eye.
* Subjects using ophthalmic medication(s) other than artificial tears for treatment of ocular pathology.
* Subjects with a history of autoimmune disease, connective tissue disease, or clinically significant atopic syndrome.
* Subjects with a history of herpes zoster or herpes simplex keratitis.
* Subjects with a history of steroid-responsive rise in intraocular pressure (IOP), or a preoperative IOP > 21 mmHg or glaucoma.
* Subjects with distorted, non-reactive, or decentered pupils.
* Subjects taking medication for the control of diabetes.
* Subjects on chronic systemic or topical corticosteroids or other immunosuppressive therapy that may affect wound healing, and any immuno-compromised subjects (use of intranasal steroids for seasonal allergies are acceptable).
* Subjects using systemic medications (e.g., amiodarone) or medications with significant ocular side effects.
* Subjects who are pregnant, or are considering becoming pregnant during the time of the study.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 412 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Uncorrected near visual acuity - operated eyes | 24 months postoperative
  Uncorrected near visual acuity at 40 cm of 20/40 or better

SECONDARY OUTCOMES:
Uncorrected near visual acuity - operated eyes | 24 months postoperative
  - Number of lines of improvement uncorrected near visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Robert K Maloney, MD, MA, Study Director — Maloney Vision Institute; Mickey Gordon, MD, Study Director — Gordon-Weiss-Schanzlin Vision Institute
Locations (11):
- United States (11):
  - Assil Eye Institute, Beverly Hills, California
  - Gordon-Weiss-Schanzlin, La Jolla, California
  - Maloney Vision Institute, Los Angeles, California
  - Stanford Eye and Laser Center, Palo Alto, California
  - Center for Sight, Sarasota, Florida
  - Kraft Eye Institute, Chicago, Illinois
  - Physicians Protocol, Greensboro, North Carolina
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Berkeley Eye and Laser Center, Houston, Texas
  - Hoopes Vision, Laser Correction Center, Draper, Utah
  - The Eye Center, Fairfax, Virginia

REFERENCES:
- See also: Website dedicated to patient recruitment (approved by WIRB on 4/3/2014). — http://www.TossYourReaders.com